CLINICAL TRIAL: NCT06347913
Title: Umblical Artery Systolic \Diastolic Ratio and Amniotic Fluid Index in Prediction of Fetal
Brief Title: Umblical Artery Systolic \Diastolic Ratio and Amniotic Fluid Index in Prediction of Fetal Outcome in Term Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sabrin Alnokrashy Mohamed, resident at obstetric and gynacology department at sohag university hospial, Sohag University
Other Study IDs: Soh-Med-24-03-09MS
Record Dates: First submitted 2024-03-11; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Umblical Artery Doppler in Term Pregnancy
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: ultrasound — Umbilical Artery Systolic/Diastolic Ratio and Amniotic Fluid Index in Prediction of Fetal Outcome in Term Pregnancies
  Other Names: umblical artery doppler in term pregnancy

SUMMARY:
Antepartum fetal surveillance is the cornerstone of management in pregnancy. [1] It is done primarily to reduce the incidence of adverse fetal outcomes. It minimizes morbidity by optimizing the timing of delivery. Fetus at risk of chronic hypoxia is identified and unnecessary interventions are avoided. However, fetal surveillance acts as a diagnostic modality to detect the influence of maternal, placental, and fetal factors on the fetus. The timely detection of morbid changes in the fetal status followed by adequate interventions to avoid death or disability is one of the most important objectives of prenatal care. [2] Tests now commonly done for antepartum fetal surveillance are nonstress test (NST), amniotic fluid index (AFI), biophysical profile, Doppler study of umbilical artery (UA), and middle cerebral artery (MCA).[3 6] However, AFI and UA Doppler velocimetry both form an essential part of the antenatal surveillance in the assessment of fetal well being. UA Doppler is a powerful tool that allows the obstetrician to follow a sequence of fetal hemodynamic events that happen in response to placental insufficiency. [7] However, several studies have reported higher sensitivities and specificities for UA Doppler ratio for prediction of fetal prognosis. [3 6] Amniotic fluid is the product of complex and dynamic fetal and placental physiologic processes. Disruption of the fine balance may result in overproduction or underproduction of fluid. Liquor adequacy often reflects the fetal status. Oligohydramnios is associated with increased perinatal loss. Furthermore, other studies indicate that UA velocimetry is a predictor of adverse outcomes in pregnancies complicated by oligohydramnios. [8,9] Thus, arterial Doppler velocimetry measurement may be useful in predicting adverse pregnancy outcomes adjunct to other antenatal surveillance tests, especially the AFI. Therefore, the present study will be done to evaluate the comparative assessment of UA ratio and AFI in predicting adverse perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* * Age of mother 18-40 years

  * Term pregnancy (37w6d -40w)
  * Singleton pregnancy

Exclusion Criteria:

* *Multiple pregnancy

  * Preterm pregnancy before 37w
  * Preeclampsia
  * IUGR
  * Diabetic
  * Congenital anomalies of fetus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: pregnant women term
Sampling Method: Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Umbilical Artery Systolic/Diastolic Ratio | 6 months
  Umblical Artery Systolic/Diastolic Ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arduini D, Rizzo G, Romanini C. Changes of pulsatility index from fetal vessels preceding the onset of late decelerations in growth-retarded fetuses. Obstet Gynecol. 1992 Apr;79(4):605-10. PMID 1553186